CLINICAL TRIAL: NCT02762188
Title: Genetic Biomarkers for the Response to Anti-VEGF (Vascular Endothelial Growth Factor).Treatment in Wet Age-related Macular Degeneration (Wet ARMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Laurence Postelmans, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-SAMBA
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: wet ARMD; VEGF; intra vitreal injections
MeSH Terms: conditions — Macular Degeneration | interventions — Genetic Association Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- wet ARMD patients (Experimental): Patients with the wet form of ARMD who receive or have received in the past anti VEGF intra vitreal injections. Diagnosis of wet ARMD is made based on clinical data-visual acuity, fundus presence of subretinal fluid and/or haemorrhage and/or hard exudates, fundus photographs -color and red free, optical coherence tomography (SD-OCT), fluorescein angiography and indocyanine green angiography showing the presence and activity of subretinal neovascularisation.
  Interventions: Device: Genotype analysis

INTERVENTIONS:
Device: Genotype analysis — After signing informed consent, a blood sample is taken and DNA extracted according to standard procedures. The samples are genotyped with the Mass Array iPlex Gold. Processing of the data is done using the previously described protocol by Lambrechts and co.
  Statistical analysis will be done to evaluate the association between the different genetic variants and the clinical outcomes collected during the standard of care follow-up for ARMD.

SUMMARY:
Age-Related Macular Degeneration (ARMD) is the most common cause of blindness in the adult population of the Western World. It affects the macula - the region of the retina most rich in photoreceptors and responsible for central vision. The ethiology of ARMD remains poorly understood. Population-based studies have demonstrated a complex ethiology, with contributions from a combination of genetic and environmental factors.

Two major forms of ARMD are clinically distinguishable: the dry and wet form. The latter represents the more aggressive clinical subgroup, and is characterized by the abnormal growth of new blood vessels (neovascularization) under the macula, thus leading to the accumulation of fluid under the retina, bleeding, progression to fibrosis, and finally loss of central vision.

The pathogenesis of this neovascularization is not fully understood, although the VEGF pathway is well known to be involved in angiogenesis and was implicated in the development of the new vessels under the macula. The VEGFs are the most specific and potent stimulators of the angiogenesis.

Molecules that bind and inactivate the VEGF have been developed for the treatment of ARMD and they are applied in ARMD clinic through intra vitreal injections.The difference seen in response to anti VEGF treatment for ARMD between the patients is suggestive for the presence of factors influencing the effect of the drug. Some of these could be genetic variants within genes involved in ARMD pathogenesis or VEGF pathway. Few associations with markers within genes previously found to be related with the pathogenesis of ARMD have been found. It remains unknown whether variants involved in the anti VEGF treatment response could influence the therapeutic outcome.

The purpose of this trial is to evaluate the association between a panel of selected polymorphic markers in the VEGF pathway and the response to therapy with anti VEGF antibody for ARMD. The hypothesis is that the individual genotype influences the response to the anti VEGF. This can lead to identification of genetic biomarkers allowing treatment individualization and optimization of the visual outcomes.

DETAILED DESCRIPTION:
Age-Related Macular Degeneration (ARMD) is the most common cause of blindness in the adult population of the Western World. It affects the macula - the region of the retina most rich in photoreceptors and responsible for central vision.

Despite this manifest importance, the ethiology of ARMD remains poorly understood. Population-based studies have demonstrated a complex ethiology, with contributions from a combination of genetic and environmental factors. Genome-wide association studies revealed the presence of loci associated with susceptibility in a wide range of genes, including genes involved in the complement system, cholesterol homeostasis, growth factor diffusion and angiogenesis. Smoking has been identified as a major environmental factor.

Two major forms of ARMD are clinically distinguishable: the dry and wet form. The latter represents the more aggressive clinical subgroup, and is characterized by the abnormal growth of new blood vessels (neovascularization) under the macula, thus leading to the accumulation of fluid under the retina, bleeding, progression to fibrosis, and finally loss of central vision.

The pathogenesis of this neovascularization is not fully understood, although the VEGF pathway is well known to be involved in angiogenesis and was implicated in the development of the new vessels under the macula. The VEGFs are the most specific and potent stimulators of the angiogenesis. VEGF-A is a 45kD glycoprotein binding to transmembrane tyrosine kinase receptors, VEGFRs, which activates a cascade of downstream factors. VEGF-A has the strongest pro-angiogenic effect in the retina by promoting proliferation, sprouting and tubing of the endothelial cells. It can bind to at least two receptors -VEGFR1 and VEGFR2, although the most of the proangiogenic activity appears to be mediated through VEGFR2. Expression of a VEGFR2 isoform that lacks both the intracellular signaling domain and the transmembrane domain, represents a soluble form of the receptor, inactivating VEGF extracellularly.

Similarly, molecules that bind and inactivate the VEGF have been developed for the treatment of ARMD and they are applied in ARMD clinic through intra vitreal injections. These include antibodies, a recombinant receptor fusion protein and a synthetic aptamer. The anti-VEGFA antibodies - ranibizumab and bevacizumab, off-label, have been associated with limited side-effects and significant therapeutic improvement, and became the standard in the treatment of the wet form of ARMD. Indeed, for example in the first clinical trials for ranibizumab, monthly injections of ranibizumab demonstrated an average gain in visual acuity of 6.6 and 10.7 ETDRS letters after 24 months. However, currently most clinical centres apply modified treatment protocols. Commonly used is an initial loading dose of three consecutive monthly injections and subsequent follow-up and administration of additional injections depending on the evolution of visual acuity, optical coherence tomography and fluorescein angiography data . 25% of the ARMD patients show significant improvement of the visual acuity, 70% maintain or show slightly increased visual acuity, and the remaining 5 percent of the patients fail to respond to the treatment and continue to loose vision.

The difference seen in response to anti VEGF treatment for ARMD between the patients is suggestive for the presence of factors influencing the effect of the drug. Some of these could be genetic variants within genes involved in ARMD pathogenesis or VEGF pathway. Few associations with markers within genes previously found to be related with the pathogenesis of ARMD have been found. It remains unknown whether variants involved in the anti VEGF treatment response could influence the therapeutic outcome.

A study demonstrated that the single nucleotide polymorphism (SNP) in VEGFR1 rs7993418 (TAC codon) form is associated to resistance to the anti VEGF therapy in carcinoma patients. This specific genotype leads to an increased expression of the VEGFR1 without changing the amino acid content of the protein. The increased VEGFR1 protein is most likely due to higher efficiency of messenger ribonucleic acid (mRNA) translation.

The purpose of this trial is to evaluate the association between a panel of selected polymorphic markers in the VEGF pathway and the response to therapy with anti VEGF antibody for ARMD. The hypothesis is that the individual genotype influences the response to the anti VEGF. This can lead to identification of genetic biomarkers allowing treatment individualization and optimization of the visual outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the wet form of ARMD who receive or have received in the past anti VEGF intra vitreal injections

Exclusion Criteria:

* Patients whi had received treatments other than anti VEGF, before the use of anti-VEGF
* Patients without follow-up
* Patients receiving anti-VEGF because of another pathology than ARMD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Snellen visual acuity test result | Baseline
  The visual acuity test is used to determine the smallest letters you can read on a standardized chart (Snellen chart).
Snellen visual acuity test result | 3 months after treatment
  The visual acuity test is used to determine the smallest letters you can read on a standardized chart (Snellen chart).
Snellen visual acuity test result | 6 months after treatment
  The visual acuity test is used to determine the smallest letters you can read on a standardized chart (Snellen chart).
Snellen visual acuity test result | 12 months after treatment
  The visual acuity test is used to determine the smallest letters you can read on a standardized chart (Snellen chart).
Number of injections received per year | 1 year
Central foveal thickness (µm) | Baseline
  Measured by optical coherence tomography (Heidelberg & Zeiss)
Central foveal thickness (µm) | 3 months after treatment
  Measured by optical coherence tomography (Heidelberg & Zeiss)
Central foveal thickness (µm) | 6 months after treatment
  Measured by optical coherence tomography (Heidelberg & Zeiss)
Central foveal thickness (µm) | 12 months after treatment
  Measured by optical coherence tomography (Heidelberg & Zeiss)
Presence of Intra Retinal Cysts (yes/no) | Baseline
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Intra Retinal Cysts (yes/no) | 3 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Intra Retinal Cysts (yes/no) | 4 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Subretinal Fluid (yes/no) | Baseline
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Subretinal Fluid (yes/no) | 3 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Subretinal Fluid (yes/no) | 4 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Pigment Epithelial Detachment (yes/no) | Baseline
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Pigment Epithelial Detachment (yes/no) | 3 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)
Presence of Pigment Epithelial Detachment (yes/no) | 4 months after treatment
  Tested by optical coherence tomography (Heidelberg & Zeiss)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Postelmans, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No